CLINICAL TRIAL: NCT01426737
Title: The Swiss Glucose Variability Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ACH02T
Record Dates: First submitted 2011-04-18; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50mg twice/d as add-on to metformin alone over 18 months compared to an add-on therapy with gliclazide 30mg max 4x/d(metformin - gliclazide).

SUMMARY:
The purpose of this study is to explore long term glucose variability of a combination therapy of metformin and vildagliptin compared to a metformin - gliclazide combination.

Multicenter, randomized, open, parallel group, Phase IV study, of 18 months duration.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged =30 -= 75 years.
2. History of type 2 diabetes for at least 6 months.
3. Patients inadequately controlled (i.e. not reaching target) with maximum tolerated doses of metformin with HbA1c of 6.5-9.0%.
4. Patients inadequately controlled (i.e. not reaching target) with maximum tolerated doses of metformin with a body mass index (BMI) of 25-40 kg/m2.
5. Patients that are currently treated with metformin, gliclazide or both but not with other glucose lowering agents.
6. Outpatient.
7. If female of childbearing potential: Will to practice reliable birth control measures [e.g., surgical sterilization, hormonal contraception, double-barrier methods (any double combination of IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)] during study treatment and for at least 28 days after completion of study medication; not lactating or pregnant; and has a documented negative pregnancy test result at baseline.

Exclusion criteria:

1. Type 1 diabetes as defined by the American Diabetes Association (ADA).
2. Type 2 diabetes currently (last 3 months) treated with insulin or glitazones.
3. Acute or chronic diseases causing tissue hypoxia such as:

   * cardiac or respiratory insufficiency
   * myocardial infarct within the last 6 months
4. Active liver disease with alanine aminotransferase (ALAT) and / or aspartate aminotransferase (ASAT) > 3 x upper limit of normal.
5. Relevant kidney disease such as :

   * serum creatinine =133 µmol/l in males and > 124 µmol/l in females
   * proteinuria > 300 mg/l
   * status post kidney transplantation
   * severe infection
   * intravascular administration of contrast medium containing iod within the last 7 days
6. Severe neuropathy (vibration perception at the base of the big toes <2/8).
7. Active proliferative diabetic retinopathy.
8. Any clinically relevant major organ system disease including mental illnesses
9. History of malignancy
10. Pancreatitis
11. Porphyria
12. Severe disturbances of the adrenal gland
13. Severe disturbances of the thyroid gland
14. Allergy to vildagliptin or one of the excipients
15. Allergy to metformin or one of the excipients
16. Allergy to gliclazide, sulfonylurea or sulfonamides or one of the excipients.
17. Drug or alcohol abuse.
18. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive pregnancy test (serum or urine).
19. Any other condition that could interfere with the participation in the study according to the study protocol or with the ability to cooperate and comply with the study procedures.
20. Treatment with any investigational drug, within 30 days or 5 half-lives before screening, whichever is longer.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Mean amplitude of glycemic excursion as described by Service et al. (1970) calculated from the glucose excursions of the CGMS profiles using MiniMedSolution Software (MedtronicMiniMed). | 48h

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Universitiy Hospital, Zurich, Switzerland